CLINICAL TRIAL: NCT00798746
Title: Role of Pyloric Drainage in Reflux Symptoms After Esophagectomy for Cancer
Brief Title: Quality of Life After Esophagectomy for Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0465
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; pyloric drainage; pyloric drainage procedure; reflux; reflux symptoms; esophagectomy; Quality of Life; Health-related quality of life; HRQL
MeSH Terms: conditions — Esophageal Neoplasms; Gastroesophageal Reflux | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pyloric Drainage Procedure: Esophagectomy with pyloric drainage procedure
  Interventions: Behavioral: Telephone Questionnaire
- No Pyloric Drainage Procedure: Esophagectomy without pyloric drainage procedure
  Interventions: Behavioral: Telephone Questionnaire

INTERVENTIONS:
Behavioral: Telephone Questionnaire — Ten questions regarding symptoms of reflux
  Other Names: Reflux Survey; Gastrointestinal Symptoms Rating Scale; GSRS; Quality of life questionnaires; Health-related quality of life; HRQL

SUMMARY:
The purpose of the current study is to assess the role of pyloric drainage procedure on altering the reflux effect on the quality of life in patients who underwent esophagectomy. Researchers hypothesize that the patients who underwent minimally invasive esophagectomies without pyloric drainage experience less reflux symptoms and therefore have a better quality of life.

DETAILED DESCRIPTION:
Surgery is considered curative for patients with esophageal cancer. The minimally invasive approach was developed such that laparoscopy and thoracoscopy replace large abdominal and thoracic incisions. For both open and minimally invasive procedures, patients have many adjustments to overcome in order to regain quality of life that is within the norm. In a recent study on the health-related quality of life (HRQL) after curative surgical resection, symptoms of reflux was the only variable that worsened with statistical significance.

The study plan is to retrospectively compare two groups of patients: those who underwent esophagectomy with pyloric drainage procedure and those who did not. The study will be done using all MD Anderson patients who underwent minimally invasive esophagectomies, in which pyloroplasty and pyloromyotomy are not standard procedures. Clinically relevant data and demographic information will be collected retrospectively for the two groups including age, gender, Body Mass Index, level of anastomosis, and time elapsed since surgery. All patients will be interviewed via telephone. At least two attempts will be made to contact each patient.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are 18 years-old or older
2. Patients who received esophagectomy indicated for primary esophageal cancer, either adenocarcinoma or squamous cell carcinoma
3. Patients who received minimally invasive or transthoracic or transhiatal or three-field esophagectomy at MDACC during or after 2004
4. Patients who are English-speaking and of any ethnicity
5. Patients with prior cancers, any clinical stage of esophageal carcinoma, any performance status (as rated by American Society of Anesthesiologist Risk Scale), received or did not receive preoperative treatment, had level of anastomosis in either neck or chest

Exclusion Criteria:

1) Patients who received esophagectomies indicated for emergency, salvage or redo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who received minimally invasive or transthoracic or transhiatal or three-field esophagectomy for primary esophageal cancer at MDACC during or after 2004.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Reflux Symptoms: Open Esophagectomy versus Minimally Invasive | Survey response collected at single point in time.
  Comparison of reflux symptoms in patients who underwent open esophagectomies with pyloric drainage and those who received minimally invasive esophagectomies without pyloric drainage. The survey consisted of ten questions regarding symptoms associated with reflux using Gastrointestinal Symptoms Rating Scale (GSRS). Responses to degree of reflux distress rated on a six-point scale for questions with "0" indicating no heartburn symptoms and "5" indicating most symptoms experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Reza J. Mehran, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org